CLINICAL TRIAL: NCT05470465
Title: Clinical Study to Investigate the Effect of Administration of Selective Serotonin Reuptake Inhibitors (SSRIs) and an Opioid on Ventilation
Brief Title: Effect of Selective Serotonin Reuptake Inhibitors (SSRIs) and an Opioid on Ventilation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Food and Drug Administration (FDA) (U.S. Federal Agency)
Collaborators: Spaulding Clinical Research LLC (Other); Leiden University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: SCR-012
Record Dates: First submitted 2022-07-14; First posted 2022-07-22 (Actual); Results first posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Hypercapnia; Ventilatory Depression
MeSH Terms: conditions — Hypercapnia; Respiratory Insufficiency | interventions — Oxycodone; Paroxetine; Escitalopram

STUDY DESIGN:
Intervention Model Description: This is a 3-period, double-blind, randomized crossover study. The duration of each treatment period will be 21 days in addition to a three-week washout between periods. The duration of study participation will be 106 days (excluding the screening period).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be double-blind, and the blind will be maintained through a randomization schedule held by the dispensing pharmacist. Treatments (escitalopram, paroxetine, or placebo) will be over-encapsulated. The pharmacist (and designated staff member responsible for confirmation of study drug dose) will be unblinded to subject treatment assignment; however, the pharmacist will not perform any study procedures other than study drug preparation and dispensing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A: Placebo (Placebo Comparator): Participants will receive placebo on days 1-21 for this treatment period. Oxycodone will be administered on days 6, 12, and 21 of this treatment period.
  Interventions: Drug: Placebo and Oxycodone
- Treatment B: Paroxetine (Experimental): Participants will receive paroxetine on days 1-21 for this treatment period. Oxycodone will be administered on days 6, 12, and 21 of this treatment period.
  Interventions: Drug: Paroxetine and Oxycodone
- Treatment C: Escitalopram (Experimental): Participants will receive escitalopram on days 1-21 for this treatment period. Oxycodone will be administered on days 6, 12, and 21 of this treatment period.
  Interventions: Drug: Escitalopram and Oxycodone

INTERVENTIONS:
Drug: Placebo and Oxycodone — Participants will receive placebo on days 1-21 for this treatment period. Oxycodone 10 mg (2 x 5 mg tablets) will be administered on days 6, 12, and 21 of this treatment period.
  Arms: Treatment A: Placebo
Drug: Paroxetine and Oxycodone — Participants will receive 40 mg paroxetine (2 x 20 mg tablets) on days 1-6 and 60 mg paroxetine (3 x 20 mg tablets) on days 7-21 for this treatment period. Oxycodone 10 mg (2 x 5 mg tablets) will be administered on days 6, 12, and 21 of this treatment period.
  Arms: Treatment B: Paroxetine
Drug: Escitalopram and Oxycodone — Participants will receive 20 mg escitalopram (2 x 10 mg tablets) on days 1-6 and 30 mg escitalopram (3 x 10 mg tablets) on days 7-21 for this treatment period. Oxycodone 10 mg (2 x 5 mg tablets) will be administered on days 6, 12, and 21 of this treatment period.
  Arms: Treatment C: Escitalopram

SUMMARY:
This study is designed to evaluate the effects of the coadministration of paroxetine or escitalopram with an opioid on ventilation. Ventilation will be assessed using a rebreathing methodology. This study will evaluate chronic and acute dosing of paroxetine and escitalopram combined with an opioid as well as chronic and acute dosing of the two drugs without coadministration of an opioid.

This study is a 3-period, randomized, placebo-controlled crossover study conducted with 25 healthy participants. Each participant will receive each of the 3 treatments (placebo/oxycodone, paroxetine/oxycodone, escitalopram/oxycodone) in a randomized order.

DETAILED DESCRIPTION:
This study is designed to evaluate the effects of the coadministration of paroxetine or escitalopram, two selective serotonin reuptake inhibitors (SSRI), with an opioid on hypercapnic ventilation. Hypercapnic ventilation will be assessed under both hyperoxic and hypoxic conditions using the Duffin rebreathing method. This method allows for critical physiological measurements and thresholds to be captured that can then be used to model the effects of drugs when there are dynamic changes in oxygen partial pressure (PO2) and carbon dioxide partial pressure (PCO2), such as during a real-world opioid overdose.

SSRIs take approximately 3 weeks to reach maximal therapeutic effect, which correlates with the time required for pre-synaptic inhibitory serotonergic receptors to desensitize. Therefore, drug-effects on ventilation should be evaluated under steady state conditions.

This study is randomized, placebo-controlled crossover study which includes three 21-day periods conducted with 25 healthy participants. Participants will receive each of the 3 treatments (placebo/oxycodone, paroxetine/oxycodone, or escitalopram/oxycodone) in a randomized order. Paroxetine dosing will range from 40-60 mg once daily (QD) and escitalopram dosing will range from 20-30 mg QD. Subjects will receive 10 mg oxycodone on three different days each period. Subjects will undergo 6 days of rebreathing and time-matched pupillary assessments along with 3 separate days of ECG assessments each period. Additionally, blood samples will be collected for determination of plasma concentrations for each study drug on days with rebreathing and ECG assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Subject signs an Institutional Review Board (IRB) approved written informed consent and privacy language as per national regulations (e.g., Health Insurance Portability and Accountability Act authorization) before any study related procedures are performed.
2. Subject is a healthy, non-smoking man or woman, 18 to 50 years of age, inclusive, who has a body mass index of 18.5 to 33.0 kg/m2, inclusive, at Screening.
3. Subject has normal medical history findings, clinical laboratory results, vital sign measurements, pulse oximetry, 12-lead ECG results, and physical examination findings at screening or, if abnormal, the abnormality is not considered clinically significant (as determined and documented by the investigator or designee).
4. Subject must have a negative test result for alcohol and drugs of abuse at screening and check-in days.
5. Subject must test negative for severe acute respiratory syndrome corona virus 2 (SARS-CoV-2) by a rapid antigen test at check-in for all study periods. If a subject's test comes back as invalid, the test can be repeated.
6. Female subjects must be of non-childbearing potential (confirmed with follicle-stimulating hormone levels > 40 milli-international unit [mIU]/mL) or, if they are of childbearing potential, they must: 1) have been strictly abstinent for 1 month before check-in (Day -1) and agree to remain strictly abstinent for the duration of the study and for at least 1month after the last application of study drug; OR 2) be practicing 2 highly effective methods of birth control (as determined by the investigator or designee; one of the methods must be a barrier technique) from at least 1 month before check-in (Day -1) until at least 1 month after the end of the study.
7. Male subjects must agree to practice 2 highly effective methods of birth control (as determined by the investigator or designee) from at least 1 month before check-in (Day -1) until at least 1 month after the last dose of study drug.
8. Subject is highly likely (as determined by the investigator) to comply with the protocol defined procedures and to complete the study.

Exclusion Criteria:

1. Subject has used any prescription or nonprescription drugs (including aspirin or NSAIDs and excluding oral contraceptives and acetaminophen) within 14 days or 5 half-lives (whichever is longer) or complementary and alternative medicines within 28 days before the first dose of study drug. This includes prescription or nonprescription ophthalmic drugs.
2. Subject is currently participating in another clinical study of an investigational drug or has been treated with any investigational drug within 30 days or 5 half-lives (whichever is longer) of the compound.
3. Subject has used nicotine-containing products (e.g., cigarettes, cigars, chewing tobacco, snuff, electronic cigarettes) within 6 weeks of Screening. Subjects must refrain from using these throughout the study.
4. Subject has consumed alcohol, xanthine containing products (e.g., tea, coffee, cola), caffeine, grapefruit, or grapefruit juice within 24 h of check-in. Subjects must refrain from ingesting these throughout the study.
5. Subject has a history or evidence of a clinically significant disorder, condition, or disease (e.g., cancer, human immunodeficiency virus [HIV], hepatic or renal impairment) that, in the opinion of the investigator would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion. This includes subjects with any underlying medical conditions that put subjects at increased risk of severe illness from coronavirus disease 2019 (COVID-19) based on the Centers for Disease Control and Prevention (CDC) guidelines.
6. Subject has any signs or symptoms at screening or check-in of any study periods that are consistent with COVID-19. Per current CDC recommendations this includes subjects with the symptoms cough or shortness of breath or difficulty breathing, or at least two of the following symptoms: fever, chills, repeated shaking with chills, muscle pain, headache, sore throat or new loss of taste/smell. In addition, the subject has any other findings suggestive of COVID-19 risk in the opinion of the investigator.
7. Subject has known or suspected allergies or sensitivities to any study drugs.
8. Subject has clinical laboratory test results (hematology, serum chemistry and urinalysis) at Screening or period check-in that are outside the reference ranges provided by the clinical laboratory and considered clinically significant by the investigator. Clinical laboratory results may be repeated once, as needed, for confirming results at Screening and period check-in.
9. Subject has a positive test result at Screening for HIV 1 or 2 antibody, hepatitis C virus antibodies, or hepatitis B surface antigen.
10. Subject is unable or unwilling to undergo multiple venipunctures for blood sample collection because of poor tolerability or poor venous access.
11. Female subject is currently pregnant or lactating or was within 3 months of before enrollment.
12. Subject has a history of opioid or psychotropic drugs within 60 days of the start of the study.
13. Subject has a history of asthma that has required medication within the last five years.
14. Subject has non-reactive or misshapen pupil(s) or damaged orbit structure or surrounding soft tissue is edematous or has an open lesion.
15. Subject has a Mallampati score of >2.
16. Subject's Duffin rebreathing data is of poor quality or subject does not agree to remain clean-shaven for all days when the Duffin rebreathing procedure is performed.
17. Subject has a history of sleep disorders, Panic disorders, Panic Attacks, Generalized Anxiety Disorder, or any associated Diagnostic and Statistical Manual of Mental Disorders diagnosis or condition.
18. Subject has a history of or currently has hypoventilation syndrome or sleep apnea and is on non-invasive ventilation.
19. Subject has a history of unexplained syncope, structural heart disease, long QT syndrome, heart failure, myocardial infarction, angina, unexplained cardiac arrhythmia, Torsades de Pointes, ventricular tachycardia, or placement of a pacemaker or implantable defibrillator. Subjects will be also excluded if there is a family history of long QT syndrome (genetically proven or suggested by sudden death of a close relative to cardiac causes at a young age) or Brugada syndrome.
20. Subject has a history of suicidal ideation or previous suicide attempts.
21. Subject has a safety 12-lead ECG result at Screening or check-in at any study period with evidence of any of the following abnormalities:

    * QTc using Fridericia correction (QTcF)>430 msec
    * PR interval>220 msec or <120msec
    * QRS duration>110 msec
    * Second- or third-degree atrioventricular block
    * Complete left or right bundle branch block or incomplete right bundle branch block
    * Heart rate <50 or >90 beats per minute
    * Pathological Q-waves (defined as Q-wave>40 msec)
    * Ventricular pre-excitation
22. Subject has a skin condition likely to compromise ECG electrode placement.
23. Any individual with breast implants.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-17 (Actual); Study Completion 2023-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Matousek, D.O., Principal Investigator — Spaulding Clinical Research LLC
Locations (1):
- Spaulding Clinical Research, West Bend, Wisconsin, United States

REFERENCES:
- [Background] Xu L, Krishna A, Stewart S, Shea K, Racz R, Weaver JL, Volpe DA, Pilli NR, Narayanasamy S, Florian J, Patel V, Matta MK, Stone MB, Zhu H, Davis MC, Strauss DG, Rouse R. Effects of sedative psychotropic drugs combined with oxycodone on respiratory depression in the rat. Clin Transl Sci. 2021 Nov;14(6):2208-2219. doi: 10.1111/cts.13080. Epub 2021 Jun 16. PMID 34080766
- [Background] Rebuck AS. Measurement of ventilatory response to CO2 by rebreathing. Chest. 1976 Jul;70(1 Suppl):118-21. doi: 10.1378/chest.70.1_supplement.118. No abstract available. PMID 939123
- [Background] van der Schrier R, Jonkman K, van Velzen M, Olofsen E, Drewes AM, Dahan A, Niesters M. An experimental study comparing the respiratory effects of tapentadol and oxycodone in healthy volunteers. Br J Anaesth. 2017 Dec 1;119(6):1169-1177. doi: 10.1093/bja/aex295. PMID 29029015
- [Background] van der Schrier R, Roozekrans M, Olofsen E, Aarts L, van Velzen M, de Jong M, Dahan A, Niesters M. Influence of Ethanol on Oxycodone-induced Respiratory Depression: A Dose-escalating Study in Young and Elderly Individuals. Anesthesiology. 2017 Mar;126(3):534-542. doi: 10.1097/ALN.0000000000001505. PMID 28170358
- [Background] Nutt DJ, Forshall S, Bell C, Rich A, Sandford J, Nash J, Argyropoulos S. Mechanisms of action of selective serotonin reuptake inhibitors in the treatment of psychiatric disorders. Eur Neuropsychopharmacol. 1999 Jul;9 Suppl 3:S81-6. doi: 10.1016/s0924-977x(99)00030-9. PMID 10523062
- [Background] Czachura JF, Rasmussen K. Effects of acute and chronic administration of fluoxetine on the activity of serotonergic neurons in the dorsal raphe nucleus of the rat. Naunyn Schmiedebergs Arch Pharmacol. 2000 Sep;362(3):266-75. doi: 10.1007/s002100000290. PMID 10997729
- [Background] Casey K, Duffin J, McAvoy GV. The effect of exercise on the central-chemoreceptor threshold in man. J Physiol. 1987 Feb;383:9-18. doi: 10.1113/jphysiol.1987.sp016392. PMID 3116207
- [Background] Duffin J, McAvoy GV. The peripheral-chemoreceptor threshold to carbon dioxide in man. J Physiol. 1988 Dec;406:15-26. doi: 10.1113/jphysiol.1988.sp017365. PMID 3151077
- [Background] Dong TW, MacLeod DB, Santoro A, Augustine Z, Barth S, Cooter M, Moon RE. A methodology to explore ventilatory chemosensitivity and opioid-induced respiratory depression risk. J Appl Physiol (1985). 2020 Sep 1;129(3):500-507. doi: 10.1152/japplphysiol.00460.2020. Epub 2020 Jul 16. PMID 32673158
- [Background] Read DJ. A clinical method for assessing the ventilatory response to carbon dioxide. Australas Ann Med. 1967 Feb;16(1):20-32. doi: 10.1111/imj.1967.16.1.20. No abstract available. PMID 6032026
- [Background] Gorman JM, Browne ST, Papp LA, Martinez J, Welkowitz L, Coplan JD, Goetz RR, Kent J, Klein DF. Effect of antipanic treatment on response to carbon dioxide. Biol Psychiatry. 1997 Dec 1;42(11):982-91. doi: 10.1016/s0006-3223(97)00160-1. PMID 9386849
- [Background] Bertani A, Perna G, Arancio C, Caldirola D, Bellodi L. Pharmacologic effect of imipramine, paroxetine, and sertraline on 35% carbon dioxide hypersensitivity in panic patients: a double-blind, random, placebo-controlled study. J Clin Psychopharmacol. 1997 Apr;17(2):97-101. doi: 10.1097/00004714-199704000-00006. PMID 10950471
- [Background] Robillard R, Saad M, Ray LB, BuJaki B, Douglass A, Lee EK, Soucy L, Spitale N, De Koninck J, Kendzerska T. Selective serotonin reuptake inhibitor use is associated with worse sleep-related breathing disturbances in individuals with depressive disorders and sleep complaints: a retrospective study. J Clin Sleep Med. 2021 Mar 1;17(3):505-513. doi: 10.5664/jcsm.8942. PMID 33118928

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Sequence ABC: Participants first received treatment A and then crossed over to the sequential treatments with three weeks of washout in between treatments.
  Treatments are as follows:
  Treatment A (Placebo and Oxycodone): Participants receive placebo on days 1-21 and Oxycodone 10 mg (2 x 5 mg tablets) on days 6, 12, and 21 of this treatment period.
  Treatment B (Paroxetine and Oxycodone): Participants receive 40 mg paroxetine (2 x 20 mg tablets) on days 1-6 and 60 mg paroxetine (3 x 20 mg tablets) on days 7-21 for this treatment period. Oxycodone 10 mg (2 x 5 mg tablets) is administered on days 6, 12, and 21 of this treatment period.
  Treatment C (Escitalopram and Oxycodone): Participants receive 20 mg escitalopram (2 x 10 mg tablets) on days 1-6 and 30 mg escitalopram (3 x 10 mg tablets) on days 7-21 for this treatment period. Oxycodone 10 mg (2 x 5 mg tablets) is administered on days 6, 12, and 21 of this treatment period.
- Treatment ACB: Participants first received treatment A and then crossed over to the sequential treatments with three weeks of washout in between treatments.
  Treatments are as follows:
  Treatment A (Placebo and Oxycodone): Participants receive placebo on days 1-21 and Oxycodone 10 mg (2 x 5 mg tablets) on days 6, 12, and 21 of this treatment period.
  Treatment C (Escitalopram and Oxycodone): Participants receive 20 mg escitalopram (2 x 10 mg tablets) on days 1-6 and 30 mg escitalopram (3 x 10 mg tablets) on days 7-21 for this treatment period. Oxycodone 10 mg (2 x 5 mg tablets) is administered on days 6, 12, and 21 of this treatment period.
  Treatment B (Paroxetine and Oxycodone): Participants receive 40 mg paroxetine (2 x 20 mg tablets) on days 1-6 and 60 mg paroxetine (3 x 20 mg tablets) on days 7-21 for this treatment period. Oxycodone 10 mg (2 x 5 mg tablets) is administered on days 6, 12, and 21 of this treatment period.
- Treatment BAC: Participants first received treatment B and then crossed over to the sequential treatments with three weeks of washout in between treatments.
  Treatments are as follows:
  Treatment B (Paroxetine and Oxycodone): Participants receive 40 mg paroxetine (2 x 20 mg tablets) on days 1-6 and 60 mg paroxetine (3 x 20 mg tablets) on days 7-21 for this treatment period. Oxycodone 10 mg (2 x 5 mg tablets) is administered on days 6, 12, and 21 of this treatment period.
  Treatment A (Placebo and Oxycodone): Participants receive placebo on days 1-21 and Oxycodone 10 mg (2 x 5 mg tablets) on days 6, 12, and 21 of this treatment period.
  Treatment C (Escitalopram and Oxycodone): Participants receive 20 mg escitalopram (2 x 10 mg tablets) on days 1-6 and 30 mg escitalopram (3 x 10 mg tablets) on days 7-21 for this treatment period. Oxycodone 10 mg (2 x 5 mg tablets) is administered on days 6, 12, and 21 of this treatment period.
- Treatment BCA: Participants first received treatment B and then crossed over to the sequential treatments with three weeks of washout in between treatments.
  Treatments are as follows:
  Treatment B (Paroxetine and Oxycodone): Participants receive 40 mg paroxetine (2 x 20 mg tablets) on days 1-6 and 60 mg paroxetine (3 x 20 mg tablets) on days 7-21 for this treatment period. Oxycodone 10 mg (2 x 5 mg tablets) is administered on days 6, 12, and 21 of this treatment period.
  Treatment C (Escitalopram and Oxycodone): Participants receive 20 mg escitalopram (2 x 10 mg tablets) on days 1-6 and 30 mg escitalopram (3 x 10 mg tablets) on days 7-21 for this treatment period. Oxycodone 10 mg (2 x 5 mg tablets) is administered on days 6, 12, and 21 of this treatment period.
  Treatment A (Placebo and Oxycodone): Participants receive placebo on days 1-21 and Oxycodone 10 mg (2 x 5 mg tablets) on days 6, 12, and 21 of this treatment period.
- Treatment CAB: Participants first received treatment C and then crossed over to the sequential treatments with three weeks of washout in between treatments.
  Treatments are as follows:
  Treatment C (Escitalopram and Oxycodone): Participants receive 20 mg escitalopram (2 x 10 mg tablets) on days 1-6 and 30 mg escitalopram (3 x 10 mg tablets) on days 7-21 for this treatment period. Oxycodone 10 mg (2 x 5 mg tablets) is administered on days 6, 12, and 21 of this treatment period.
  Treatment A (Placebo and Oxycodone): Participants receive placebo on days 1-21 and Oxycodone 10 mg (2 x 5 mg tablets) on days 6, 12, and 21 of this treatment period.
  Treatment B (Paroxetine and Oxycodone): Participants receive 40 mg paroxetine (2 x 20 mg tablets) on days 1-6 and 60 mg paroxetine (3 x 20 mg tablets) on days 7-21 for this treatment period. Oxycodone 10 mg (2 x 5 mg tablets) is administered on days 6, 12, and 21 of this treatment period.
- Treatment CBA: Participants first received treatment C and then crossed over to the sequential treatments with three weeks of washout in between treatments.
  Treatments are as follows:
  Treatment C (Escitalopram and Oxycodone): Participants receive 20 mg escitalopram (2 x 10 mg tablets) on days 1-6 and 30 mg escitalopram (3 x 10 mg tablets) on days 7-21 for this treatment period. Oxycodone 10 mg (2 x 5 mg tablets) is administered on days 6, 12, and 21 of this treatment period.
  Treatment B (Paroxetine and Oxycodone): Participants receive 40 mg paroxetine (2 x 20 mg tablets) on days 1-6 and 60 mg paroxetine (3 x 20 mg tablets) on days 7-21 for this treatment period. Oxycodone 10 mg (2 x 5 mg tablets) is administered on days 6, 12, and 21 of this treatment period.
  Treatment A (Placebo and Oxycodone): Participants receive placebo on days 1-21 and Oxycodone 10 mg (2 x 5 mg tablets) on days 6, 12, and 21 of this treatment period.
Period: Overall Study
Arm/Group | Treatment Sequence ABC | Treatment ACB | Treatment BAC | Treatment BCA | Treatment CAB | Treatment CBA
Started | 5 | 4 | 5 | 5 | 4 | 4
Completed | 4 | 4 | 2 | 4 | 4 | 4
Not Completed | 1 | 0 | 3 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Participants received a treatment in a randomized order and then crossed over to the sequential treatments with three weeks of washout in between treatments.
  Treatments are as follows:
  Treatment A (Placebo and Oxycodone): Participants receive placebo on days 1-21 and Oxycodone 10 mg (2 x 5 mg tablets) on days 6, 12, and 21 of this treatment period.
  Treatment B (Paroxetine and Oxycodone): Participants receive 40 mg paroxetine (2 x 20 mg tablets) on days 1-6 and 60 mg paroxetine (3 x 20 mg tablets) on days 7-21 for this treatment period. Oxycodone 10 mg (2 x 5 mg tablets) is administered on days 6, 12, and 21 of this treatment period.
  Treatment C (Escitalopram and Oxycodone): Participants receive 20 mg escitalopram (2 x 10 mg tablets) on days 1-6 and 30 mg escitalopram (3 x 10 mg tablets) on days 7-21 for this treatment period. Oxycodone 10 mg (2 x 5 mg tablets) is administered on days 6, 12, and 21 of this treatment period.
Arm/Group | Total
Number analyzed (Participants) | 27
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36 [31 to 40.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 18
  More than one race | 0
  Unknown or Not Reported | 2
Body Weight [Median (Inter-Quartile Range); unit: kg] | 77 [66 to 84]
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m2] | 24.4 [22.8 to 27.5]
Minute Ventilation [Median (Inter-Quartile Range); unit: L/min] | 9.4 [8.7 to 10.1]
Respiratory Rate [Median (Inter-Quartile Range); unit: breaths/min] | 13.6 [12.0 to 15.2]
Tidal Volume [Median (Inter-Quartile Range); unit: L] | 0.79 [0.66 to 0.92]
End-tidal Carbon Dioxide [Median (Inter-Quartile Range); unit: mmHg] | 36.0 [33.9 to 38.1]
Oxygen Saturation [Median (Inter-Quartile Range); unit: percentage] | 96.8 [95.9 to 97.7]

OUTCOME MEASURES:

1. Primary Outcome: Minute Ventilation at 55mm Hg End Tidal CO2 (VE55) Under Hyperoxic Conditions on Day 21
Description: Comparison of escitalopram or paroxetine with oxycodone to oxycodone alone. Rebreathing data will be analyzed by regression of the minute ventilation versus partial pressure of end tidal CO2 (PETCO2) data to estimate VE55. Resulting VE55 data will be compared using a linear mixed effects model. Comparison will be at 5 hours on day 21.
Time Frame: 5 hours on day 21
Measure: Mean (95% Confidence Interval); unit: L/min
Groups:
- Paroxetine + Oxycodone: Participants will receive 40 mg paroxetine (2 x 20 mg tablets) on days 1-6 and 60 mg paroxetine (3 x 20 mg tablets) on days 7-21 for this treatment period. Oxycodone 10 mg (2 x 5 mg tablets) will be administered on days 6, 12, and 21 of this treatment period.
- Escitalopram + Oxycodone: Participants will receive 20 mg escitalopram (2 x 10 mg tablets) on days 1-6 and 30 mg escitalopram (3 x 10 mg tablets) on days 7-21 for this treatment period. Oxycodone 10 mg (2 x 5 mg tablets) will be administered on days 6, 12, and 21 of this treatment period.
- Placebo + Oxycodone: Participants will receive placebo on days 1-21 for this treatment period. Oxycodone 10 mg (2 x 5 mg tablets) will be administered on days 6, 12, and 21 of this treatment period.
Arm/Group | Paroxetine + Oxycodone | Escitalopram + Oxycodone | Placebo + Oxycodone
Number analyzed (Participants) | 22 | 22 | 22
L/min | 20.2 [15.8 to 24.6] | 21.2 [16.8 to 25.6] | 26.7 [22.3 to 31.2]
Statistical Analysis 1: Comparison: Paroxetine + Oxycodone vs Placebo + Oxycodone; Sample size and power were calculated based on 2 primary outcomes (day 20 and day 21) with adjustment for multiplicity (α=.025). The assessments with paroxetine or escitalopram were considered as separate experiments. A sample size of 20 participants was determined to have 90 percent power at a 1-sided significance level to detect a 4 L/min decrease in the primary end point (ventilation at 55 mmHg end-tidal carbon dioxide) assuming a standard deviation of 5 L/min; Test type: Superiority; p < 0.001, Mixed Models Analysis — To demonstrate an effect of oxycodone with paroxetine compared to oxycodone alone, it is necessary that the upper bound of the one-sided 97.5% confidence interval (CI) in the least-square mean VE55 difference between treatments < 0 L/min; The Kenward-Roger approximation will be used to estimate denominator degrees of freedom for tests of fixed effects; Mean Difference (Final Values) = -6.5, 97.5% CI 1-sided [upper limit -3.1] — Comparison was the effect of oxycodone and paroxetine compared to oxycodone and placebo
Statistical Analysis 2: Comparison: Escitalopram + Oxycodone vs Placebo + Oxycodone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.001, Mixed Models Analysis — To demonstrate an effect of oxycodone with escitalopram compared to oxycodone alone, it is necessary that the upper bound of the one-sided 97.5% confidence interval (CI) in the least-square mean VE55 difference between treatments < 0 L/min; The Kenward-Roger approximation will be used to estimate denominator degrees of freedom for tests of fixed effects; Mean Difference (Final Values) = -5.5, 97.5% CI 1-sided [upper limit -2.1] — Comparison was the effect of oxycodone and escitalopram compared to oxycodone and placebo

2. Primary Outcome: VE55 Under Hyperoxic Conditions on Day 20
Description: Comparison of escitalopram or paroxetine to placebo. Rebreathing data will be analyzed by regression of the minute ventilation versus partial pressure of end tidal CO2 (PETCO2) data to estimate VE55. Resulting VE55 data will be compared using a linear mixed effects model. Comparison will be at 5 hours on day 20.
Time Frame: 5 hours on day 20
Measure: Mean (95% Confidence Interval); unit: L/min
Groups:
- Paroxetine: Participants will receive 40 mg paroxetine (2 x 20 mg tablets) on days 1-6 and 60 mg paroxetine (3 x 20 mg tablets) on days 7-21 for this treatment period. Oxycodone 10 mg (2 x 5 mg tablets) will be administered on days 6, 12, and 21 of this treatment period.
- Escitalopram: Participants will receive 20 mg escitalopram (2 x 10 mg tablets) on days 1-6 and 30 mg escitalopram (3 x 10 mg tablets) on days 7-21 for this treatment period. Oxycodone 10 mg (2 x 5 mg tablets) will be administered on days 6, 12, and 21 of this treatment period.
- Placebo: Participants will receive placebo on days 1-21 for this treatment period. Oxycodone 10 mg (2 x 5 mg tablets) will be administered on days 6, 12, and 21 of this treatment period.
Arm/Group | Paroxetine | Escitalopram | Placebo
Number analyzed (Participants) | 22 | 22 | 22
L/min | 30.8 [25.9 to 35.7] | 30.4 [25.5 to 35.3] | 37.4 [32.4 to 42.3]
Statistical Analysis 1: Comparison: Paroxetine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.002, Mixed Models Analysis — To demonstrate an effect of paroxetine compared to placebo, it is necessary that the upper bound of the one-sided 97.5% confidence interval (CI) in the least-square mean VE55 difference between treatments < 0 L/min; The Kenward-Roger approximation will be used to estimate denominator degrees of freedom for tests of fixed effects; Mean Difference (Final Values) = -6.5, 97.5% CI 1-sided [upper limit -2.1] — Comparison was the effect of paroxetine compared to placebo
Statistical Analysis 2: Comparison: Escitalopram vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.003, Mixed Models Analysis — To demonstrate an effect of escitalopram compared to placebo, it is necessary that the upper bound of the one-sided 97.5% confidence interval (CI) in the least-square mean VE55 difference between treatments < 0 L/min; The Kenward-Roger approximation will be used to estimate denominator degrees of freedom for tests of fixed effects; Mean Difference (Final Values) = -6.9, 97.5% CI 1-sided [upper limit -2.5] — Comparison was the effect of escitalopram compared to placebo

3. Secondary Outcome: VE55 Under Hyperoxic Conditions on Day 6
Description: Comparison of escitalopram or paroxetine with oxycodone to oxycodone alone. Rebreathing data will be analyzed by regression of the minute ventilation versus partial pressure of end tidal CO2 (PETCO2) data to estimate VE55. Resulting VE55 data will be compared using a linear mixed effects model. Comparison will be at 5 hours on day 6.
Time Frame: 5 hours on day 6
Measure: Mean (95% Confidence Interval); unit: L/min
Arm/Group | Paroxetine + Oxycodone | Escitalopram + Oxycodone | Placebo + Oxycodone
Number analyzed (Participants) | 22 | 22 | 22
L/min | 18.5 [14.8 to 22.2] | 20.0 [16.4 to 23.7] | 25.6 [21.8 to 29.4]
Statistical Analysis 1: Comparison: Paroxetine + Oxycodone vs Placebo + Oxycodone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis — Secondary analyses are not adjusted for multiplicity. To demonstrate an effect of oxycodone and paroxetine compared to oxycodone, the upper bound of the one-sided 97.5% CI in the least-square mean VE55 difference between treatments < 0 L/min; The Kenward-Roger approximation will be used to estimate denominator degrees of freedom for tests of fixed effects; Mean Difference (Final Values) = -7.1, 97.5% CI 1-sided [upper limit -4.1] — Comparison was the effect of oxycodone and paroxetine compared to oxycodone and placebo at day 6 at 5 hours
Statistical Analysis 2: Comparison: Escitalopram + Oxycodone vs Placebo + Oxycodone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis — Secondary analyses are not adjusted for multiplicity. To demonstrate an effect of oxycodone and escitalopram compared to oxycodone, the upper bound of the one-sided 97.5% CI in the least-square mean VE55 difference between treatments < 0 L/min; The Kenward-Roger approximation will be used to estimate denominator degrees of freedom for tests of fixed effects; Mean Difference (Final Values) = -5.6, 97.5% CI 1-sided [upper limit -2.6] — Comparison was the effect of oxycodone and escitalopram compared to oxycodone and placebo at day 6 at 5 hours

4. Secondary Outcome: VE55 Under Hyperoxic Conditions on Day 12
Description: Comparison of escitalopram or paroxetine with oxycodone to oxycodone alone. Rebreathing data will be analyzed by regression of the minute ventilation versus partial pressure of end tidal CO2 (PETCO2) data to estimate VE55. Resulting VE55 data will be compared using a linear mixed effects model. Comparison will be at 5 hours on day 12.
Time Frame: 5 hours on day 12
Measure: Mean (95% Confidence Interval); unit: L/min
Arm/Group | Paroxetine + Oxycodone | Escitalopram + Oxycodone | Placebo + Oxycodone
Number analyzed (Participants) | 22 | 22 | 22
L/min | 18.1 [14.0 to 22.3] | 21.4 [17.3 to 25.5] | 28.2 [24.0 to 32.4]
Statistical Analysis 1: Comparison: Paroxetine + Oxycodone vs Placebo + Oxycodone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; The Kenward-Roger approximation will be used to estimate denominator degrees of freedom for tests of fixed effects; Mean Difference (Final Values) = -10.1, 97.5% CI 1-sided [upper limit -5.9] — Comparison was the effect of oxycodone and paroxetine compared to oxycodone and placebo at day 12 at 5 hours
Statistical Analysis 2: Comparison: Escitalopram + Oxycodone vs Placebo + Oxycodone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.003, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 2]; The Kenward-Roger approximation will be used to estimate denominator degrees of freedom for tests of fixed effects; Mean Difference (Final Values) = -6.9, 97.5% CI 1-sided [upper limit -2.7] — Comparison was the effect of oxycodone and paroxetine compared to oxycodone and placebo at day 12 at 5 hours

5. Secondary Outcome: VE55 Under Hyperoxic Conditions on Day 5
Description: Comparison of escitalopram or paroxetine to placebo. Rebreathing data will be analyzed by regression of the minute ventilation versus partial pressure of end tidal CO2 (PETCO2) data to estimate VE55. Resulting VE55 data will be compared using a linear mixed effects model. Comparison will be at 5 hours on day 5.
Time Frame: 5 hours on day 5
Measure: Mean (95% Confidence Interval); unit: L/min
Arm/Group | Paroxetine | Escitalopram | Placebo
Number analyzed (Participants) | 22 | 22 | 22
L/min | 31.1 [26.8 to 35.4] | 28.6 [24.3 to 32.9] | 42.6 [38.3 to 46.9]
Statistical Analysis 1: Comparison: Paroxetine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis — Secondary analyses are not adjusted for multiplicity. To demonstrate an effect of paroxetine compared to placebo, the upper bound of the one-sided 97.5% CI in the least-square mean VE55 difference between treatments < 0 L/min; The Kenward-Roger approximation will be used to estimate denominator degrees of freedom for tests of fixed effects; Mean Difference (Final Values) = -11.6, 97.5% CI 1-sided [upper limit -6.5] — Comparison was the effect of paroxetine compared to placebo at day 5 at 5 hours
Statistical Analysis 2: Comparison: Escitalopram vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis — Secondary analyses are not adjusted for multiplicity. To demonstrate an effect of escitalopram compared to placebo, the upper bound of the one-sided 97.5% CI in the least-square mean VE55 difference between treatments < 0 L/min; The Kenward-Roger approximation will be used to estimate denominator degrees of freedom for tests of fixed effects; Mean Difference (Final Values) = -14.0, 97.5% CI 1-sided [upper limit -9.0] — Comparison was the effect of escitalopram compared to placebo at day 5 at 5 hours

6. Secondary Outcome: VE55 Under Hyperoxic Conditions on Day 11
Description: Comparison of escitalopram or paroxetine to placebo. Rebreathing data will be analyzed by regression of the minute ventilation versus partial pressure of end tidal CO2 (PETCO2) data to estimate VE55. Resulting VE55 data will be compared using a linear mixed effects model. Comparison will be at 5 hours on day 11.
Time Frame: 5 hours on day 11
Measure: Mean (95% Confidence Interval); unit: L/min
Arm/Group | Paroxetine | Escitalopram | Placebo
Number analyzed (Participants) | 22 | 22 | 22
L/min | 27.3 [21.8 to 32.9] | 32.0 [26.4 to 37.5] | 41.4 [35.8 to 47.0]
Statistical Analysis 1: Comparison: Paroxetine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]; The Kenward-Roger approximation will be used to estimate denominator degrees of freedom for tests of fixed effects; Mean Difference (Final Values) = -14.1, 97.5% CI 1-sided [upper limit -8.5] — Comparison was the effect of paroxetine compared to placebo at day 11 at 5 hours
Statistical Analysis 2: Comparison: Escitalopram vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 2]; The Kenward-Roger approximation will be used to estimate denominator degrees of freedom for tests of fixed effects; Mean Difference (Final Values) = -9.5, 97.5% CI 1-sided [upper limit -3.8] — Comparison was the effect of escitalopram compared to placebo at day 11 at 5 hours

ADVERSE EVENTS:
Time Frame: 106 days
Arm/Group | Treatment A: Placebo | Treatment B: Paroxetine | Treatment C: Escitalopram
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 26/27 | 26/27 | 26/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A: Placebo (N=27) | Treatment B: Paroxetine (N=27) | Treatment C: Escitalopram (N=27)
Nausea (Gastrointestinal disorders) | 6 (13) | 4 (4) | 6 (6)
Dizziness (Nervous system disorders) | 5 (5) | 4 (4) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 7 (7) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 4 (4) | 1 (1)
Drowsiness (Nervous system disorders) | 4 (4) | 2 (2) | 2 (2)
Application site irritation (General disorders) | 3 (3) | 2 (2) | 2 (2)
Insomnia (Nervous system disorders) | 1 (1) | 4 (4) | 1 (1)
Infusion site bruising (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 1 (1)
Contusion (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Brain fog (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1) | 1 (1)
Vision blurred (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Vessel puncture site bruise (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Vessel puncture site erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 2 (3)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Infusion site pain (General disorders) | 2 (2) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Change in bowel habit (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Vessel puncture site pain (General disorders) | 1 (2) | 0 (0) | 0 (0)
Infusion site erythema (General disorders) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Anorgasmia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep talking (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Paroncychia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Diffuse alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Burns first degree (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal Pruritis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Euphoric mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Irritability (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hot Flush (General disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperacusis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
A limitation of this study was that the breathing assessments were conducted in a controlled experimental setting with healthy volunteers which may not be representative of actual at-risk individuals having an overdose. However, the methods used provide a safe way to assess ventilatory effects of drugs as carbon dioxide levels increase, which reflects the physiology of severe respiratory depression.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/65/NCT05470465/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/65/NCT05470465/SAP_001.pdf
  • Informed Consent Form (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT05470465/ICF_002.pdf